CLINICAL TRIAL: NCT04327050
Title: Prospective Clinical Trial of Magnetic Anchoring Guided Endoscopic Submucosal Dissection for Early Gastric Caner
Brief Title: Magnetic Anchoring Guided Endoscopic Submucosal Dissection for Early Gastric Caner
Acronym: MAGESD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-2017ZD1-09
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer
Keywords: magnetic anchored guidance; early gastric cancer; endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Masking Description: No masking required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic-ESD (Experimental): Patients in MAG arm will be treated using magnetic anchored guided endoscopic submucosal dissection.
  Interventions: Procedure: Magnetic anchored guided endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Magnetic anchored guided endoscopic submucosal dissection — Using magnetic anchoring technology, the magnetic pulling unit is anchored to the abdominal wall, and micro surgical tweezers are used. The tumor tissue is pulled indirectly, so that the mucosa is lifted up, which is beneficial to the peeling of the submucosa.

SUMMARY:
This study uses magnetic anchored guidance system to treat early gastric cancer by endoscopic mucosal dissection to test the advantages of magnetically anchored guidance system for surgical field exposure during endoscopic mucosal dissection.

DETAILED DESCRIPTION:
Gastric cancer is the second most common malignant tumor in China, with the highest mortality rate among all types of malignant tumors. Surgical resection is still the most effective treatment for gastric cancer. Minimally invasive surgery breaks the traditional surgical concept that the laparotomy must be performed by laparotomy. It can complete the operation that required a large incision with minimal incision trauma, and has the advantages of less trauma, faster recovery and fewer complications. At present, the application of gastroscopy and laparoscopy for early gastric cancer has reached consensus at home and abroad. Endoscopic mucosal resection of early gastric cancer is suitable for patients with intramucosal cancer and no lymph node metastasis. However, the unclear exposure of the surgical field during the operation causes difficulty in operation or conversion to open surgery is a difficult problem facing this technique. The project designed a magnetic pulling unit that can be connected through an endoscope, including external abdominal magnets, internal abdominal magnets, connecting hooks, and micro surgical tweezers. Using magnetic anchoring technology, the magnetic pulling unit is anchored to the abdominal wall, and micro surgical tweezers are used. The tumor tissue is pulled indirectly, so that the mucosa is lifted up, which is beneficial to the peeling of the submucosa. This method increases the operating space of the main hand of the endoscope, and at the same time, the magnetic clamp is used to connect the clamps so that they can move in all directions, so as to achieve the desired traction of the tumor tissue site, fully expose the surgical field, and facilitate surgical anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed as of gastric cancer by a preliminary endoscopy or biopsy sampling

Exclusion Criteria:

* Patients with a cardiac pacemaker or severe cardiac and/or pulmonary diseases
* Patients without informed consent
* Patients with other malignant tumors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
success rate | through study completion, an average of 1 year
  The rate of the complete resection of gastric lesion by magnetic anchored guided endoscopic submucosal dissection

SECONDARY OUTCOMES:
complications | measured at the time of the end of each ESD; up to 1 hour
  the complications in magnetic anchored guided endoscopic submucosal dissection

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Shuixiang He, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No